CLINICAL TRIAL: NCT01544738
Title: Aponeurotic Stimulation Effect on Parkinson Bradykinesia
Brief Title: Sensory Stimulation Effect on Movement Speed in Patients With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); Belgium: Belgian Federal Science Policy Office (BELSPO) (Unknown)
Responsible Party: Principal Investigator, Ana Bengoetxea, Assistant Professor, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LMNB-01
Record Dates: First submitted 2012-02-23; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; sensory stimulation; Bradykinesia
MeSH Terms: conditions — Parkinson Disease; Hypokinesia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Aponeurotic stimulation group (Experimental): The stimulation consisted of manipulating, with a hook (the diacutaneous fibrolysis method), the aponeurotic tissues enrobing the heads of the trunk and upper limb muscles.
  Interventions: Other: Aponeurotic stimulation (the diacutaneous fibrolysis method)
- Placebo stimulation group (Active Comparator): Placebo stimulation (PS) consisted of manipulating the skin along the same paths over the trunk, shoulder and arm muscles that were the targets for treatment in the Aponeurotic stimulation group.
  Interventions: Other: Placebo stimulation

INTERVENTIONS:
Other: Aponeurotic stimulation (the diacutaneous fibrolysis method) — Treatment consisted of manipulating, with a hook, the aponeurotic tissues enrobing the heads of the upper-limb muscles. The manipulation consisted of back and forth mobilization, applied perpendicularly to the axis of the muscular fibers. The mobilization is performed with both hands; the therapist's non-dominant hand performs a manual mobilization whereas the dominant hand follows the movement with the hook. The hook allows the therapist to be very precise about the location of the tissues that are stretched. This stretch is realized at the level of the aponeurotic fibers presenting the greatest resistance to perpendicular movement. The shape of the hook is chosen to avoid discomfort or pain during manipulation. To spread the pressure exerted by the spatula on a very local point, it is important to fill completely the curved part of the hook with the adjacent soft tissues. We manipulated muscle from the proximal insertion towards the distal, giving special attention to the tendons.
  Arms: Aponeurotic stimulation group
Other: Placebo stimulation — Placebo stimulation (PS) consisted of manipulating the skin along the same paths over the trunk, shoulder and arm muscles that were the targets for treatment in the AS group
  Arms: Placebo stimulation group

SUMMARY:
Movement slowness (bradykinesia) is one of the main motor symptoms in Parkinson Disease (PD). Several studies have shown that patients with PD exhibit slowness because they are unable to modulate, in an optimal way, the velocity of voluntary motor acts not induced by external stimulation. Indeed, these patients have difficulties to integrate multi-sensorial information, mainly proprioception.

The investigators investigated changes in shoulder velocity during pointing movements by patients with PD after stimulation of soft tissues (aponeurosis) of upper limb muscles. The stimulation consisted of manipulating, with a hook (the diacutaneous fibrolysis method), the aponeurotic tissues enrobing the heads of the upper limb muscles. This technique has previously been shown to decrease passive tension and the tendon reflex response of the manipulated muscle group. The investigators hypothesis is that aponeurotic manipulation of shoulder muscles therefore creates a modification in the proprioceptive information, which in return temporarily decreases the bradykinesia of shoulder movements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson Disease

Exclusion Criteria:

* Patients with a limitation in the shoulder range of motion necessary to perform pointing movements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
3D kinematic movement parameters and upper limb muscles electromyographic activation | Participants will be followed for the duration of the clinical test (2 weeks)

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | Participants will be followed for the duration of the clinical test (2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Bengoetxea, PhD, Principal Investigator — Université Libre de Bruxelles; Françoise Leurs, PhD Student, Study Chair — Université Libre de Bruxelles; Leslie Rigal, Master Student, Study Chair — Université Libre de Bruxelles; Guy Cheron, PhD, Study Director — Université Libre de Bruxelles
Locations (1):
- ULB-FSM Laboratory of neurophysiology and movement biomechanics, Brussels, Belgium